CLINICAL TRIAL: NCT01715350
Title: A Phase 2 Clinical Study to Explore the Optimal Dosage/Administration of PM012 Tablet in Alzheimer's Disease: Double-Blind, Randomized Between Placebo Control Group and Dose Groups, Parallel-Design, Multicenter Study
Brief Title: Study to Explore the Optimal Dosage/Administration in Alzheimer's Disease
Acronym: ADD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VTBIO Co. LTD (Industry)
Collaborators: ADM Korea Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PM012-P2
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Placebo Comparator): • Drug : Placebo 2 tablet
  The drug will be taken with water within 30 minutes after breakfast and supper. Even if no meal is taken, dosing will not be omitted and the drug should be taken with enough amount of water.
  Interventions: Drug: Placebo
- Dose group 1 (Experimental): * Drug : Placebo 1 tablet + Study drug 1 tablet
  * Study drug(650-mg PM012 tablet)
  The drug will be taken with water within 30 minutes after breakfast and supper. Even if no meal is taken, dosing will not be omitted and the drug should be taken with enough amount of water.
  Interventions: Drug: PM012; Drug: Placebo
- Dose group 2 (Experimental): * Drug : Study drug 2 tablet
  * Study drug (650-mg PM012 tablet)
  The drug will be taken with water within 30 minutes after breakfast and supper. Even if no meal is taken, dosing will not be omitted and the drug should be taken with enough amount of water.
  Interventions: Drug: PM012

INTERVENTIONS:
Drug: PM012 — * The drug will be taken with water within 30 minutes after breakfast and supper.
  * 650mg/1 tablet, PO, 12weeks
  Other Names: 650-mg PM012 tablet
  Arms: Dose group 1; Dose group 2
Drug: Placebo — * The drug will be taken with water within 30 minutes after breakfast and supper.
  * 650mg/1 tablet, PO, 12weeks
  Other Names: Placebo (for PM012)
  Arms: Dose group 1; Placebo group

SUMMARY:
The investigators intend to perform exploratory evaluation of the treatment effectiveness and safety of PM012 Tablet of PuriMED Co., Ltd. at 2 doses in Korean patients with mild to moderate dementia of Alzheimer's type. To achieve this, this study aims to compare each dose with placebo control for the efficacy and safety to explore the clinically optimal dose of PM012 Tablet for therapeutic confirmatory (phase 3) clinical studies.

DETAILED DESCRIPTION:
1. Period of study

   -48 months from the date of KFDA approval of the protocol
2. Study subjects

   -Patients with mild to moderate Alzheimer's disease
3. Study objectives

   1. Primary objective

      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on cognitive effect assessed by ADAS-cog at Week 12 post-dose
   2. Secondary objectives

      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on cognitive effect assessed by ADAS-cog at Week 8 post-dose
      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on overall functional effect assessed by CDR at Weeks 8 and 12 post-dose
      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on activities of daily living assessed by K-IADL at Weeks 8 and 12 post-dose
      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on behavioral changes assessed by NPI at Weeks 8 and 12 post-dose
      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on cognitive effect assessed by K-MMSE at Weeks 8 and 12 post-dose
      * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on improvement on VAS assessed by Senile Dementia Pattern Identification Diagnosis System at Weeks 8 and 12 post-dose
4. Study drug / Comparator

   -650-mg PM012 Tablet by PuriMED Co., Ltd. / Placebo
5. Dosage/ Administration and Method of administration

   1. Placebo group

      * Morning:Placebo 2T, Evening:Placebo 2T
   2. Dose group 1

      * Morning:Placebo 1T+Study drug 1T, Evening:Placebo 1T+Study drug 1T
   3. Dose group 2

      * Morning:Study drug 2T, Evening:Study drug 2T
   4. Study drug is 650-mg PM012 tablet
   5. The drug will be taken with water within 30 minutes after breakfast and supper.
   6. Even if no meal is taken, dosing will not be omitted and the drug should be taken with enough amount of water.
6. Treatment duration

   -12 weeks
7. Number of subjects

   1. placebo group

      * Efficacy population:42, Drop-out(20%)included:53
   2. Dose group 1

      * Efficacy population:42, Drop-out(20%)included:53
   3. Dose group 2

      * Efficacy population:42, Drop-out(20%)included:53
   4. Total

      * Efficacy population:126, Drop-out(20%)included:159
8. Study method

   * This study is designed to be a multicenter, randomized, double-blind, parallel placebo group and 2 dose groups, phase 2 clinical study in patients with dementia of Alzheimer's type aged ≥ 50 and ≤ 85 years.
   * Once a subject voluntarily provides the written consent to participate in the study, he/she will be randomized only if meeting the inclusion criteria and exclusion criteria through screening test. Randomized subjects will receive the study drug or the placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1)Male and female patients aged ≥ 50 and ≤ 85 years
* 2)Clinically diagnosed with probable Alzheimer's disease based on DSM-IV and NINCDS-ADRDA criteria
* 3)K-MMSE score of 12~26 at screening visit
* 4)For females: 2 years of confirmed menopause or surgical sterilization.
* 5)Able to walk (including the use of aids)
* 6)Able to perform procedures for cognitive and other tests
* 7)Residing with a life-long guardian willing to accompany the subject's on all visits, oversee his/her compliance with the procedures specified in the protocol and the study drug, and report his/her condition.
* 8)Having signed him/herself or his/her legally acceptable representative having signed the written informed consent form

Exclusion Criteria:

* 1)Possible, probable, or definite vascular dementia by NINDS-AIREN criteria
* 2)History and/or evidence (result of CT or MRI performed within the past 12 months or at screening) of other CNS disease (cerebrovascular disease, structural or developmental anomaly, epilepsy, contagious, degenerative or infectious/demyelinating CNS condition) as a cause of dementia
* 3)Delusion, delirium, epilepsy and other neurological pathology on neurological examination
* 4)Abnormal test result on vitamin B12, syphilis serology, and thyroid stimulating hormone (TSH) tests that are thought to contribute to the subject's dementia severity or be a cause of dementia
* 5)History of significant psychiatric disease such as schizophrenia or bipolar affective disorder that may interfere with the participation in this study in the opinion of the investigator, or current depression (GDS ≥ 18)
* 6)Past history of known or suspected seizures including febrile convulsion, unexplained recent unconsciousness or past history of significant head trauma with unconsciousness.
* 7)Gastrointestinal, endocrine and cardiovascular disease not controlled by diet or pharmacologic therapy
* 8)Cardiac disease such as myocardial infarction or valvular disease of heart, arrhythmia within 3 months of the study start
* 9)Diabetes mellitus not controlled by hypoglycemic agent or insulin-dependent diabetes mellitus
* 10)Past history of alcohol or other drug abuse
* 11)Having taken acetylcholinesterase inhibitor or memantine within the past 3 months
* 12)Hypertension with systolic blood pressure of > 165 mmHg or diastolic blood pressure of > 96 mmHg
* 13)Severe renal impairment (serum creatinine ≥ 1.7 mg/dl)
* 14)Severe hepatic impairment (ALT, AST, or bilirubin ≥ 2.0 x upper limit of normal)
* 15)Is taking or expected to take disallowed concomitant medication
* 16)History of clinically significant drug hypersensitivity
* 17)Is ineligible to participate in this study in the judgment of the investigator

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
ADAS-cog | Week 12 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on cognitive effect assessed by ADAS-cog at Week 12 post-dose

SECONDARY OUTCOMES:
ADAS-cog | Weeks 8 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on cognitive effect assessed by ADAS-cog at Week 8 post-dose
CDR | Weeks 8 and 12 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on overall functional effect assessed by CDR at Weeks 8 and 12 post-dose
K-IADL | Weeks 8 and 12 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on activities of daily living assessed by K-IADL at Weeks 8 and 12 post-dose
NPI | Weeks 8 and 12 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on behavioral changes assessed by NPI at Weeks 8 and 12 post-dose
K-MMSE | Weeks 8 and 12 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on cognitive effect assessed by K-MMSE at Weeks 8 and 12 post-dose
VAS | at Weeks 8 and 12 post-dose
  * To compare the efficacy of 2 doses of PM012 Tablet and placebo based on improvement on VAS assessed by Senile Dementia Pattern Identification Diagnosis System at Weeks 8 and 12 post-dose
AE | while the subject is receiving the treatment
  * To compare the safety based on treatment-emergent adverse events, laboratory tests (hematology/blood chemistry, urinalysis), physical examination, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Seoung-Hun Cho, M.D., Principal Investigator — Kyung Hee University Oriental Medicine Hospital; Chang-Uk Lee, M.D., Principal Investigator — The Catholic University of Korea; Hyun-Kook Lim, M.D., Principal Investigator — Saint Vincent's Hospital, Korea; Jun-Hong Lee, M.D., Principal Investigator — National Health Insurance Service Ilsan Hospital
Locations (4):
- South Korea (4):
  - Kyung Hee University Oriental Medicine Hospital, Seoul, Dongdaemun-gu
  - National Health Insurance Corporation Ilsan Hospital, Goyang, Ilsandong-gu
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Paldal-gu
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seocho-gu

REFERENCES:
- See also: Korea Food & Drug Administration — http://www.kfda.go.kr